CLINICAL TRIAL: NCT01725711
Title: Osseointegrated Prostheses for the Rehabilitation of Amputees.
Acronym: OPRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrum (Industry)
Collaborators: Sahlgrenska University Hospital (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R402-98
Record Dates: First submitted 2012-10-15; First posted 2012-11-14 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Transfemoral Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implant System (Experimental)
  Interventions: Device: OPRA Implant System

INTERVENTIONS:
Device: OPRA Implant System

SUMMARY:
Patients with transfemoral amputations (TFA) frequently experience problems related to the use of socket-suspended prostheses 1-3. These problems increase with short or deformed stumps 4. The potential for improvement is substantial. Based on the very good long-term results with osseointegrated titanium implants for edentulous patients 5, osseointegrated hearing aids 6, cranio-facial prostheses 7 and prostheses for thumb-amputated patients 8, the clinical development of osseointegrated prostheses for TFA started in 1990, in Gothenburg, Sweden. The concept has gradually been modified and improved. In 1999, a prospective clinical trial began.

The hypothesis is that the treatment will improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Transfemoral amputation

Exclusion Criteria:

* Transfemoral amputation due to vascular disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1999-05; Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Q-TFA Prosthetic Use Score | 0,1,2,3,5,7,10,15,20 years
  The primary efficacy variable is the change in Q-TFA Prosthetic Use Score as compared baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, VG, Sweden